CLINICAL TRIAL: NCT04260386
Title: A Study to Assess the Utility of a New Proforma in Simulated Clinical Scenarios of Maternal Cardiac Arrest
Brief Title: Assessing a New Proforma for Maternal Cardiac Arrest
Status: Terminated | Type: Observational
Why Stopped: The study closed early due to COVID-19
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W19/004; 264325 (Other: Integrated Research Application System)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Maternal Death; Cardiac Arrest; Heart Arrest
Keywords: Maternal Cardiac Arrest; Clinical Scenarios Simulation
MeSH Terms: conditions — Maternal Death; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Staff receiving the MOMS training: Delegates taking part in the routine Multidisciplinary Obstetric and Midwifery Simulation (MOMS) training course at the Chelsea and Westminster Hospital.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — During the cardiac arrest scenario, the delegates observing will be asked to refer to the maternal cardiac arrest proforma and record those details of events that they are able to see/hear from the video link. In addition, the proforma will be provided to the team taking part in the simulation. One or more team members would routinely be given the role of 'scribe', recording events as they occur. The proforma is accompanied by explanatory notes on how to use it.
  Delegates (observers plus scribes) will then be asked to complete a questionnaire, seeking their opinions on the usefulness of the proforma. Questionnaires will be linked to the written consent forms by a participant ID number.

SUMMARY:
During the Multidisciplinary Obstetric and Midwifery Simulation (MOMS) course, groups of delegates manage simulated clinical emergencies, whilst the remaining delegates observe the scenario via a video link.

The delegates observing the cardiac arrest scenario will be asked to refer to the proforma and record those details of events that they are able to see/hear from the video link. In addition, the proforma will be provided to the team taking part in the simulation. Delegates (observers plus scribes) will then be asked to complete a questionnaire seeking their opinions on the usefulness of the proforma.

DETAILED DESCRIPTION:
The use of standardised proformas can improve the quality and completeness of data collection in healthcare settings. In a previous study we have found that medical records examined by the Confidential Enquiries into Maternal Deaths (CEMD) 2009-2012 were variable in their quality, often poor and in need of improvement. In view of this, we have developed a proforma to assist the quality of record-keeping during maternal cardiac arrest, using a modified Delphi process amongst a multidisciplinary group of CEMD assessors. The present application is for a study evaluating clinicians' views of this proforma and its usefulness in a simulator setting (as maternal cardiac arrest is so rare, evaluation in actual cases would be a very lengthy and expensive venture; such a study would have to be multicentre and would require a preliminary evaluation such as the one being proposed here, anyway).

One hundred participants will take part in the study during the routine Multidisciplinary Obstetric and Midwifery Simulation (MOMS) training course at the Chelsea and Westminster Hospital. During the course, groups of delegates manage simulated clinical emergencies, whilst the remaining delegates observe the scenario via a video link. A brief information sheet and explanation will be provided before consent is sought to take part in the study.

During the cardiac arrest scenario, the delegates observing will be asked to refer to the proforma and record those details of events that they are able to see/hear from the video link. In addition, the proforma will be provided to the team taking part in the simulation. One or more team members would routinely be given the role of 'scribe', recording events as they occur. Delegates (observers plus scribes) will then be asked to complete a questionnaire seeking their opinions on the usefulness of the proforma. All of the data will be collected pseudo-anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Delegates taking part in the routine Multidisciplinary Obstetric and Midwifery Simulation training course at the Chelsea and Westminster Hospital.

Exclusion Criteria:

* Unwillingness to participate and provide written consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One hundred participants will take part in the study during the routine Multidisciplinary Obstetric and Midwifery Simulation (MOMS) training course at the Chelsea and Westminster Hospital. During the course, groups of delegates manage simulated clinical emergencies, whilst the remaining delegates observe the scenario via a video link.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Views of the multidisciplinary team members on the utility of the proforma in simulated clinical scenarios of maternal cardiac arrest. | Each participant is expected to be in the study for one day.
  The primary outcome is the views of multidisciplinary team members on the usefulness of the maternal cardiac arrest proforma. Researchers will not be assessing the completion of the proforma so they will not be collecting these at the end of the simulation. They have chosen to test the proforma during simulated maternal cardiac arrest, as the best practicable surrogate for an actual maternal cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Roderick, BMBCh BA, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel A, Rockall A, Guthrie A, Gleeson F, Worthy S, Grubnic S, Burling D, Allen C, Padhani A, Carey B, Cavanagh P, Peake MD, Brown G. Can the completeness of radiological cancer staging reports be improved using proforma reporting? A prospective multicentre non-blinded interventional study across 21 centres in the UK. BMJ Open. 2018 Oct 2;8(10):e018499. doi: 10.1136/bmjopen-2017-018499. PMID 30282676
- [Background] Green AR, Hoyle J, Knight MK, Yentis SM. Documentation of maternal cardiac arrest in clinical case notes. International Journal of Obstetric Anesthesia 2017; 31 Suppl 1: S41.
- [Background] A proforma for recording maternal cardiac arrest, R Soysa, MK Knight, SM Yentis. International Journal of Obstetric Anesthesia 2019 (in press).